CLINICAL TRIAL: NCT01131468
Title: The Evaluation of the Protective Effect of N-Acetylcysteine Against Drug Induced Ototoxicity in Peritoneal Dialysis Patients
Brief Title: Prevention of Drug Induced Ototoxicity in Peritoneal Dialysis Patients by N-Acetylcysteine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: TC Erciyes University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OTOTOXICITY RESEARCH IN PD
Record Dates: First submitted 2010-05-17; First posted 2010-05-27 (Estimated); Last update posted 2010-05-27 (Estimated); Status verified 2010-03

CONDITIONS: Drug-induced Ototoxicity in Peritoneal Dialysis Patients
Keywords: ototoxicity; aminoglycoside; vancomycine; peritoneal dialysis; peritonitis
MeSH Terms: conditions — Ototoxicity; Peritonitis | interventions — Acetylcysteine

ARMS (2):
- N-acetylcysteine (Experimental): N-acetylcysteine 600 mg twice daily + vancomycine and/or amikacin
  Interventions: Drug: N-acetylcysteine
- Controls (No Intervention): Vancomycine and/or amikacin alone
  Interventions: Drug: N-acetylcysteine

INTERVENTIONS:
Drug: N-acetylcysteine — N-acetylcysteine 600 mg twice daily or vancomycine+amikacin alone

SUMMARY:
The purpose of this study is to determine whether N-acetylcysteine is effective in the prevention of hearing loss in both ears due to aminoglycoside and/or vancomycine induced ototoxicity in peritoneal dialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* End-stage renal disease
* Undergoing continuous ambulatory peritoneal dialysis as a renal replacement therapy
* Clinical diagnosis of a peritonitis episode in a continuous ambulatory peritoneal dialysis patient
* Developing the first continuous ambulatory peritoneal dialysis related peritonitis episode

Exclusion Criteria:

* Being treated with aminoglycoside antibiotics and vancomycine within the previous 3 months
* Detection of mechanical occlusion of external ear
* Having signs of disturbed integrity of tympanic membrane on otoscopy or tympanometry
* History of a continuous ambulatory peritoneal dialysis related peritonitis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-02; Primary Completion 2010-04 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bulent Tokgoz, MD, Principal Investigator — Erciyes University School of Medicine
Locations (1):
- Erciyes University School of Medicine Department of Nephrology, Kayseri, Turkey (Türkiye)

REFERENCES:
- [Derived] Tokgoz B, Ucar C, Kocyigit I, Somdas M, Unal A, Vural A, Sipahioglu M, Oymak O, Utas C. Protective effect of N-acetylcysteine from drug-induced ototoxicity in uraemic patients with CAPD peritonitis. Nephrol Dial Transplant. 2011 Dec;26(12):4073-8. doi: 10.1093/ndt/gfr211. Epub 2011 May 6. PMID 21551083